CLINICAL TRIAL: NCT06215495
Title: A Novel Target Delineation Scheme Based on RTOG(Radiation Therapy Oncology Group) and EORTC(European Organisation for Research and Treatment of Cancer) Guidelines Impact on Survival Time and Radiotherapy Complications in High-grade Glioma Patients: a Single-center Randomized Single-blind Clinical Trial
Brief Title: A Novel Target Delineation Scheme in High-grade Glioma Patients: a Randomized Single-blind Clinical Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zhujiang Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-KY-010-01
Record Dates: First submitted 2023-10-30; First posted 2024-01-22 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-01

CONDITIONS: Radiation Toxicity; MRI Simulated Positioning; High Grade Glioma; Progression-free Survival; Overall Survival
MeSH Terms: conditions — Radiation Injuries; Glioma

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- reduced CTV (clinical target volume) and PTV (planning target volume) (Experimental)
  Interventions: Radiation: reduced target volume
- EORTC CTV (clinical target volume) and PTV (planning target volume) (Active Comparator)
  Interventions: Radiation: EORTC (European organisation for research and treatment of cancer) target volume

INTERVENTIONS:
Radiation: reduced target volume — Delineate residual tumor(GTVp) and tumor bed(GTVtb) on enhanced contrast CT-MRI(T2 fluid attenuated inversion recovery, T2 FLAIR) fusion images. GTVtb and GTVp are expanded by 1cm to CTV_6000.
  The clinical target volume_6000 cGy (CTV_6000) is partially reduced beyond the skull and midline. According to the CT-MRI(T2 FLAIR) fusion images, the edema area that cannot be seen on contrast-enhanced CT and only can be seen on MRI should be included.
  If CTV_6000 includes thalamus, basal ganglia, brainstem or motor cortex, dose of these areas will be limited no more than 54Gy
  Arms: reduced CTV (clinical target volume) and PTV (planning target volume)
Radiation: EORTC (European organisation for research and treatment of cancer) target volume — delineate according to EORTC guideline
  Arms: EORTC CTV (clinical target volume) and PTV (planning target volume)

SUMMARY:
The main question it aims to answer are:

1. whether the new target delineation scheme can improve Progression-free Survival
2. whether it can reduce the incidence of radiation complications in high-grade glioma patients.

Participants in trial group will be performed radiotherapy of new target delineation method after the completion of the operation within 4-6 weeks., while participants in the control group be performed radiotherapy of EORTC(European organisation for research and treatment of cancer) target delineation method.Temozolomide 75 mg / ( m² · d ) will be given to both groups of patients during radiotherapy. After radiotherapy, its dose changes to 150 ~ 200 mg / ( m² · d ) for 5 days and stopped for 23 days as a cycle. There are 6 cycles in total.

ELIGIBILITY:
Inclusion Criteria:

1. High-grade glioma (2021 WHO grade III or IV)
2. Age between 18-65 years old, Karnofsky performance status (KPS) score ≥ 70
3. result of pregnancy test being negative within 7 days before enrollment, only applicable to women with reproductive potential
4. The patient voluntarily joined this study and signed an informed consent form
5. Willing to return for follow-up
6. Willing to provide tissue and blood samples for this research
7. Surgical treatment was completed without any postoperative complications (such as consciousness disorders, hematomas, lung infection and cardiac insufficiency)
8. Radiotherapy within 4-6 weeks after surgery
9. No contraindications for taking temozolomide

Exclusion Criteria:

1. Low-grade glioma(2021 WHO grade I or II)
2. had or having other type of malignant cancers
3. not having been performed gross total resection of tumor
4. Severe active comorbidities, systemic diseases or other serious comorbidities that would render the patient unsuitable for participation in this study or seriously interfere with the appropriate evaluation of the safety and toxicity of the prescribed regimen in the judgment of the investigator, including but not limited to persistent or active infections, symptomatic congestive heart failure, unstable angina pectoris, arrhythmia, or mental illness；
5. Baseline MRI indicates a previous or recent risk of cerebral hemorrhage or hernia;
6. Pregnancy or lactation, or pregnancy or childbirth during the expected trial period(from pre-screening or screening visits until 120 days after the last trial treatment)
7. Unable to perform brain magnetic resonance imaging;
8. Allergic to CT contrast agent, unable to perform enhanced CT examination;
9. Remote transfer;
10. Medical contraindications for receiving radiation therapy, such as active systemic lupus or scleroderma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2024-02-18 (Actual); Primary Completion 2027-05-28 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
progression-free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 3 years
  confirm if the participant's cancer progresses or he/she dies every time back to the hospital during screening and follow-up

SECONDARY OUTCOMES:
overall survival | From date of randomization until the date of death from any cause, assessed up to 3 year
  confirm if the participant dies every time back to the hospital during screening and follow-up
European organisation for research and treatment of cancer QLQ-C30 (EORTC-QLQ-C30) | through study completion, up to 3 years
  EORTC-QLQ-C30 questionnaire
radiotherapy complication incidence | through study completion, up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Yujing Tan, Doctor, Principal Investigator — +8613560347303
Locations (1):
- southern medical university affiliated Zhujiang Hospital, Guangzhou, China